CLINICAL TRIAL: NCT06883513
Title: Osteopathic Manipulative Therapy(OMT) Effects on Post-Acute Sequalae of COVID-19(PASC)
Brief Title: Osteopathic Manipulative Therapy Effects on Post-Acute Sequelae of COVID-19 (PASC) or Long COVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Michael Stenta, Co-Investigator, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB Number: 23.0718
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Long-COVID; PASC; Long COVID Syndrome
Keywords: Long-COVID; PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OMT treatment (Experimental): Participants will undergo OMT protocol that has been shown to improve Long-COVID smell intensity
  Interventions: Other: Osteopathic Manipulative Therapy Long-COVID protocol; Other: Osteopathic Manipulative Therapy NOT Long-COVID treatment protocol
- OMT sham (Sham Comparator): Participants will undergo an OMT treatment sequence that is not targeting areas that was targeted by the OMT treatment group. This will still be OMT, just not Long-COVID targeted OMT. Individuals who have had OMT before study will still be receiving treatment so they will be "blinded".
  Interventions: Other: Osteopathic Manipulative Therapy NOT Long-COVID treatment protocol

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy Long-COVID protocol — 1. Rib Raising
  2. Suboccipital Release
  3. Thoracic Inlet Release
  4. Miller Pump
  5. Pedal Pump
  6. Suboccipital Release
  7. Cranial Sequence of Sinus Effleurage followed by indirect force within vault hold
  Other Names: Osteopathic Manipulative Medicine
  Arms: OMT treatment
Other: Osteopathic Manipulative Therapy NOT Long-COVID treatment protocol — 1. Bilateral Trapezius Direct Myofascial Release
  2. Still's technique of the First rib Bilaterally:
  3. Hamstring Muscle Energy

SUMMARY:
This study is investigating the effects of using an Osteopathic Manipulative Therapy (OMT) treatment protocol that was shown to statistically improve smell in individuals suffering from Long-COVID olfactory (smell) dysfunction in a small single-blinded pilot trial conducted during 2021.

The questions this study is trying to answer are:

1. Does this OMT protocol improve other non-smell related Long-COVID symptoms
2. Do 2 OMT treatments improve Long-COVID symptoms more than 1 OMT treatment

Participants will:

1. Week 1: Take an digital survey regarding their Long-COVID symptoms undergo Long-COVID OMT treatment or a placebo treatment
2. Week 2: Take an digital survey regarding their Long-COVID symptoms then all will undergo Long-COVID OMT treatment
3. Week 3: Take an digital survey regarding their Long-COVID symptoms
4. Week 8: Take an digital survey regarding their Long-COVID symptoms

DETAILED DESCRIPTION:
II. Description of the protocol and hypothesis with pilot data:

To date, individuals suffering from Long-COVID still do not have a specific proven treatment for this disease as a whole; however, an OMT sequence that was generated for prolonged post-COVID olfactory dysfunction was shown to generate significant increase in smell intensity after one treatment. Below is the abstract for a pilot trial:

Osteopathic Manipulative Therapy Effects on Prolonged Post-COVID Olfactory Dysfunction In 2019, the emergence of SARS-CoV2 created countless threats to public health that were unique to the pathogen. One of the first cardinal symptoms of infection is a sudden loss of smell and taste. Most people who survive their infection regain their sense of smell; however, a small amount of the population have prolonged decrease, complete absence, or abnormalities of smell long after the infection has resolved. This study represents a single-blinded pilot trial conducted during 2021 to examine the effects of a single treatment with OMT in individuals who have self-identified prolonged post-COVID anosmia, hyposmia or parosmia (n=20). This study was conducted at 2 locations within Ohio University.

Patients were randomly assigned to either the OMT group or a placebo/light touch/sham group by a flip of the coin and subsequently underwent pre-treatment smell testing of 4 items (Orange, Red Onion, Bourbon, and Perfume) they were then treated based on group selection, and subsequently underwent post-treatment smell testing to determine change in olfactory function. It was hypothesized that the OMT group would have a greater improvement in olfactory function when compared to the placebo group. A Mann-Whitney test indicated that the post and pre-treatment differences in the correct smell intensity scores of red onions were significantly higher for participants who received OMT treatment (Mdn = 2.00) compared to participants who received a non-osteopathic treatment (Mdn=1.00), U=20, p=0.019, r=5. There was a correlation of an increase in smell intensity in 2 out of the 3 remaining smell items, the mean difference between pre-smell treatment and post-smell treatment in the OMT group was higher than the placebo group. This therapy is a potential treatment for individuals suffering from this PASC related symptom and should be investigated further to determine the magnitude of OMT's effects on prolonged post-COVID olfactory dysfunction.

Side effects from the treatment group in the above study were minor but included light-headedness, drowsiness. After one treatment, there was significant improvement in olfactory dysfunction in participants in the treatment group as outlined by the study above. A poster presentation for the above study was accepted at 3 national conferences (American Academy of Osteopathy, American Academy of Physical Medicine and Rehabilitation, and American College of Physicians in San Diego) this past year.

The OMT sequence generated for the above trial is reproducible and safe. The OMT protocol designed for the above trial was as follows:

1. Rib Raising: A patient sits on edge of a treatment table, the physician faces the patient and places hands on the posterior aspect of the thorax (focus of palpation being on the vertebral-chondral junction), following patient inspiration and expiration the physician elevated and depresses the rib cage in tandem. This is classically hypothesized to engage the Sympathetic chain and cause an initial stimulation followed by a decrease in sympathetic tone via decreasing restriction of the anatomical space.
2. Suboccipital Release: The patient lies supine. The physician places the pads of their phalanges slightly inferior to the occiput and then applies a slight therapeutic force to the area to stimulate CN-X. The physician stops applying pressure when a "release" of the fascial plane is appreciated by the physician. This is classically hypothesized to engage the parasympathetic nervous system and stabilize parasympathetic tone via decreasing restriction of the anatomical space.
3. Thoracic Inlet Release: The patient lies supine. The physician places each hand on the ipsilateral aspect of the thoracic inlet and then engages the anatomical space in three different planes of motions (Flexion/extension, Lateralization(Rt)/Lateralization (Lt), and Rotation(Clockwise/counterclockwise)). Once the physician engages all planes, they then place the thoracic aperture into restriction in relations to the above planes of motion and hold the position until there is a "release" or an increase in pulse of the carotids which implies a fascial plane changing to a state of decrease tone. This is classically hypothesized to decrease restriction to flow in which it relates to the thoracic inlet for lymphatic drainage.
4. Miller Pump: The patient lies supine. The physician places each hand on the ipsilateral ribs 2-4 on the anterior aspect of the thorax. The patient is instructed to inhale and exhale through their mouth. On exhalation the physician places a force into the thorax to slightly compress the thorax. During the inhalation phase of the respiratory cycle the physician maintains pressure to prevent the rib cage from expanding. On the following exhalation phase, the physician applies force to the thorax to "take up slack" that the thorax would physiologically generate on the following inhalation motion. The physician then repeats 2-3 more times pending on the patient's compliance of the physician introduced force/thorax restriction. On the following inhalation, the physician releases the force and the thorax rebounds to physiological range of motion. This is classically hypothesized to generate a negative pressure gradient that generates a rebound thoracic expansion that correlates to an influx of lymphatic drainage within the thoracic cavity via the thoracic inlet.
5. Pedal Pump: The patient lies supine. The physician places each hand on the dorsum of the patient's feet and moves the feet into dorsi-flexion followed by plantar flexion 3 times. This is classically hypothesized to assist with venous pooling in the lower extremity and "pump" venous flow as well as lymphatic flow into the greater circulation.
6. Suboccipital Release: This is repeated as this was part of the initial protocol. It is unethical to not include this step as individuals who benefitted from the initial protocol underwent this repeat maneuver and received symptomatic relief from prolonged post-COVID olfactory dysfunction. This stage is also hypothesized to continually stimulate the parasympathetic nervous symptom through re-engagement of the vagus nerve as listed above.
7. Cranial Sequence of Sinus Effleurage followed by indirect force within vault hold: This is the final aspect and hypothetically the most important aspect of the sequence. The description of this protocol will be divided in two parts (the actions required to complete and the experimental hypothesis that differentiates the classical hypothesis)

<!-- -->

1. The patient lies supine. The physician places the pads of their phalanges overtop of the lambdoid suture. The physician then applies a slight therapeutic force on the suture until a "release" of the fascial plane is appreciated by the physician. A "release" is sometimes felt as an increase in pulsatile activity. The physician then places the pads of their phalanges just lateral to the posterior-aspect of the sagittal suture until a "release" of the fascial plane is appreciated by the physician. The physician then places the pads of their contralateral thumbs just lateral to the posterior-aspect of the sagittal suture and spreads the fascia abutting the suture laterally until a "release" of the fascial plane is appreciated by the physician. The physician then places the pads of their phalanges just lateral to the midline of the frontal bone to apply a slight therapeutic spreading force until a "release" of the fascial plane is appreciated by the physician. The physician then engages the skull in the "vault hold" in which the 5th digit of each hand is overlying the ipsilateral squamous aspect of the occiput, the 4th digit is overlying the mastoid process of the temporal bones, the 3rd digit is overlying the zygomatic process of the temporal bones, the 2nd digit is overlying the greater wings of the sphenoid and the 1st digit is overlying the cranium. The physician then holds this position lightly until the cranial respiratory motion (the phenomenon of paired skull bones motion along suture lines) is appreciated. This allows the physician to determine how the sphenoid is moving relative to the occiput and parietal bones, depending on the motion that is appreciated, the physician moves the structures to the least amount of restriction and moves the bones back to their physiological baseline of which a "release" is appreciated.
2. The vault hold is classically hypothesized to be sensing the "pulse" of CSF movement as it moves through the CNS. This is where the hypothesis that is used in this study differentiates from the classical hypothesis.

   * The classical hypothesis seems incorrect. CSF is produced and consumed in "steady state". The choroid plexus generates CSF as a continuous function and arachnoid granulations absorb CSF in a continuous function. There is no "pump" as there is with the heart to generate forward blood flow. The real question is, what is generating the paired skull bones movement along suture lines, and why did this maneuver help improve olfactory function?
   * This research team is hypothesizing that this pulse appreciated on paired cranial bones on suture lines could be a pulse of the sympathetic nervous system. This is not proven, nor is it described in classical Osteopathic or Allopathic literature. This hypothesis is supported more in-depth below.

The original pilot study was designed to engage the olfactory region and correlated lymphatic and vascular drainage. Below is a brief discussion of the hypothesis for the pilot study:

The pathology of SARS-CoV-2 viral particles has been studied extensively; however, there are still speculations regarding how the virus causes a prolonged olfactory dysfunction. There is significant evidence that the SARS-CoV-2 viral particle has a spike protein (S2) that gains entrance to the human host via attaching Angiotensin-Converting-Enzyme 2 (ACE-2) receptor and is endocytosed into the cell in respiratory epithelium. It has also been determined that the Transmembrane Serine Protease Gene 2 (TMPRSS2) gene is also responsible for viral entry into the host [1]. The ACE-2 receptor and TMPRSS2 are distributed in high concentration throughout the nasal respiratory tract [1],[2].

In general, there are 4 main hypothesized mechanisms surrounding SARS-CoV-2 olfactory dysfunction:

1. general nasal obstruction due to rhinorrhea
2. olfactory neuron destruction
3. viral CNS infiltration affecting olfactory neurons
4. injury to support cells within the nasal epithelium [3].

A significant number of individuals who were infected with SARS-CoV-2 and have olfactory dysfunction do not report rhinorrhea or nasal congestion [4]. The timeline of recovery from anosmia does not align with the timeline for regeneration of olfactory neurons and support cells, causing this hypothesis to be less likely [3]. In addition, the CNS infiltration via entrance through olfactory neurons has limited evidence based on the lack of brain tissue alteration observed via magnetic resonance imaging [3].

Injury to the support cells has increasing evidence as the most likely mechanism of action in SARS-CoV-2 causing olfactory dysfunction. These support cells have significant TMPRSS2 and ACE-2 receptor expression as discussed above. It has been shown that the infection of the golden Syrian hamster with SARS-CoV-2 has shown significant damage to olfactory epithelium (OE). Bryche, et al. determined that the damages to the OE were due to significant infection of a large proportion of the sustentacular cells (OE support cells) and that there was no viral load detected within the olfactory bulb itself. They also observed significant inflammation within the sustentacular cells that they determined to be a potential cause of the OE desquamation. [5]

The pilot trial proceeded with the hypothesis that significant inflammation caused by SARS-CoV-2 damages the sustentacular cells and OE, causing prolonged olfactory dysfunction. Inflammation causes cytokine release to recruit immune cells and to fight off invading pathogens. This inflammation can be prolonged if there is not adequate blood flow to or from the inflamed area. Cytokine release causes immune cell recruitment which releases more cytokines and stimulates a chain reaction of inflammation. This positive feedback loop generates excellent recruitment of immune cells and is the basis for the body's successful immune response. Inadequate clearing of immune cells and cytokines could potentially continue this positive feedback loop long after the pathogen has been cleared.

The olfactory zone is relatively small as well as the vasculature related to it. Due to the significant inflammation caused by SARS-CoV-2 infection, it was hypothesized that the reason individuals have prolonged olfactory dysfunction is due to inadequate drainage and clearing of inflammation. The vascular and lymphatic drainage associated with sustentacular cells are not being cleared of inflammation and cellular debris, which in turn continues to contribute to individuals' prolonged olfactory dysfunction.

The research team used Osteopathic Manipulative Therapy (OMT) in an attempt to increase venous and lymphatic drainage from the olfactory region to rid the system of the positive feedback loop. OMT is a minimally invasive treatment modality that is currently in use for a variety of ailments. When being done by an experienced physician, there are minimal side effects and the therapeutic effects are felt by the patient in a relatively short time period. OMT has been shown to increase lymphatic drainage [6] as well as hypothesized to increase venous sinus drainage of the cranium and more importantly stimulate cavernous sinus drainage which is responsible for a significant amount of the olfactory region's venous return. By using OMT, the physician can alter the fluid mechanics of this fluid static region and allow the olfactory area to re-establish the sense of smell.

After the conclusion of the original pilot study and evidence that the therapy offered benefit; others who were suffering with other Long-COVID symptoms requested the above OMT sequence and had subjective improvement of other non-olfactory symptoms. It was quite surprising to find these individuals would regain function and have a decrease in symptoms related to long-COVID even though the treatment sequence was designed to target the olfactory zone to reduce a positive feedback loop of inflammation.

This anecdotal evidence of individuals having improvement in function related to other long-COVID symptoms with the same protocol that was targeted to treat olfactory dysfunction suggests the hypothesis of why this OMT treatment protocol works should change. Although the treatment protocol used in the original pilot study is designed to improve lymph and vascular drainage, there could be another effect the treatment protocol is having on the body resulting in decrease in Long-COVID symptom burden.

SARS-CoV-2 infection is notorious for causing widespread sympathetic hyperactivity. In the early stages of the pandemic, individuals who were in critical condition succumbed to Acute Respiratory Distress Syndrome (ARDS). It is thought that the pathophysiology behind ARDS is related to sympathetic hyperactivity following an insult. This sympathetic hyperactivity generates "leaky" capillaries that cause extravasation of lymph to fight infection. In ARDS this increase in vascular wall permeability leads to lymph filling the viscera and inhibiting lung compliance and gas exchange which in turn generates respiratory failure.

This hypothesis has changed in regard to why people get relief from this OMT sequence and therefore the pathophysiology of Long COVID. Although there is likely a component of residual inflammation in the body related to a fluid mechanics model, anecdotal evidence would suggest a stronger driving force is leading to Long COVID symptoms. Could prolonged sympathetic hyperactivity be the root-cause of Long COVID?

This treatment protocol could generate a significant decrease in sympathetic tone quickly as well as improve lymphatic and vascular flow. This would explain why participants in the original pilot study had a significant increase in smell only 10 minutes after the treatment. This hypothesis would also explain why others treated with the sequence had a significant improvement in their non-related olfactory symptoms within 10 minutes of one treatment.

III. Trial Design:

The clinical trial design is a modified cross over study performed over an 8-week period to assess the effects of OMT on Long-COVID. This study would evaluate individuals with Long-COVID symptom burden through The Symptom Burden Questionnaire™ for Long COVID (SBQ™-LC) [7] which is to be taken before treatment. SBQ™-LC is a validated tool generated to assess for Long-COVID symptom burden generated by the University of Birmingham in the UK. A user license has been granted to the research team to utilize the SBQ™-LC. This user license allows the research team to electronically design and implement this survey independently, this will be done through Red-Cap.

In addition to the survey, the research team will acquire blood pressure (BP) and heart rate (HR) from all participants before and after treatment, as a proxy measurement of sympathetic activity. BP and HR are elevated in increased sympathetic tone states and therefore could be a relative measurement of sympathetic tone in a non-invasive and low risk manner.

There will be 2 groups: an OMT group (experimental) and a sham-OMT/placebo group (control). The control group will receive an OMT treatment that is not designed to stimulate the sympathetic nervous system, but is designed to make participants feel that they have received OMT which they will. The sham/placebo treatment regiment is listed below. The experimental group will receive the therapeutic OMT treatment as listed above. Participants will be placed into respective groups via randomization software or coinflip if software is unavailable. after completing their consent form.

The experimental group will receive OMT on week 1 and week 2. The control group will receive the sham-OMT for 1 week and then will receive OMT for 1 week. This design will allow comparison of treatment vs no treatment as well as 1 treatment vs 2 consecutive treatments.

This trial will have participants complete SBQ™-LC a total of 4 times. The 1st being upon consent and prior to any treatment (baseline). The 2nd being upon arrival for the second treatment (7 days after the first treatment). The 3rd being 7 days after their second treatment. The 4th survey will be 8 weeks post initial treatment. Goal is N=20. Based on median effect size of initial pilot data, using a treatment group and an control/sham group, the median observed effect size was 1.2 leading to an ideal n=8 per group, followed by an approximate 20% attrition rate will give n=10 per group which is a total of N=20.

The primary endpoint for this study will be the 8-week mark post initial treatment.

The OMT-Sham treatment is listed below:

1. Bilateral Trapezius Direct Myofascial Release

   a. Patient is lying supine with physician seated at the head of the bed. The physician places 2-3 digits on the superior aspect of the trapezius and engages with slight pressure until the fascial layer is engarged. Next the physician moves the fascia while maintaning enough pressure to ensure there is no slippage of the dermis in contact with the physician's finger pads and moves the myofascial plane in 3 planes of motion (Superior/inferior, Lateral/medial, and clockwise/counterclockwise rotation) the physician will then determine which of the 3 directions are restricted to movement, the physician will then engage all planes of motion into the restriction until a release is palpated.
2. Still's technique of the First rib Bilaterally:

   a. Patient is lying supine with physician standing on the side of the rib being treated. The physician grasps the forearm on the side of the rib being treated while placing the physician's other hand over the posterolateral aspect of the rib in question at the T1/Rib 1 costal articulation. The physician positions the patient's arm anteriorly and adducted. Then the physician will lift the arm into flexion and abduction in a circumduction motion, continuing the motion with the arm posterior (behind the trunk) and then back down to the side of the patient.
3. Hamstring Muscle Energy

   1. Patient lies supine. Physician stands on the same side that is being treated. The hip is flexed and knee extended to the point of the restriction. The physician will hold the leg in this position and will ask the patient to flex their knee and extend their hip while the physician resists this force for 3-5 seconds. The patient will then relax, and the physician will "take up the slack" by slightly increasing the hip flexion and knee extension. Repeat this 3 times. Have patient relax and gently set their leg back on the table.

      IIIa. Inclusion and Exclusion criteria: As with any research this is difficult, especially in the setting of Long-COVID. To date there are no official diagnostic criteria for Long-COVID or the Post-Acute Sequlae of COVID-19. It is a diagnosis of exclusion and comes from a pertinent medical history and signs and symptoms presented by an individual suffering from this ailment.

      In the light of above, the following is inclusion and exclusion criteria:

      - Individuals must claim they have had a prior positive SARS-CoV-2 test at least 6-weeks before the consenting process to proceed with the study

      - Individuals must claim they have at least one of the following symptoms greater than 6-weeks post infection that is affecting their daily life(these symptoms correlate with the SBQ™-LC):

      Table II: Symptoms of Long Covid Inclusion Criteria:

      Shortness of breath or Difficulty Breathing Difficulty with Movement (balance or tremor) Muscle Pain or stiffness Changes in sexual desire Worsening Generalized Pain Difficulty with Sleep Changes in Mood (anxiety or depression) Changes in Erectile function (Biological males only) Palpations (irregular heart beats) Altered Taste Changes in your Hair Changes in urination Dizziness Altered Smell Changes in Skin Changes in bowels Fatigue Indigestion Dry or irritated eyes Changes in sweating Difficulty with Cognition (memory or thinking) Stomach Pain Changes in menstruation (Biological females only) Chills or shivering

      - If anyone denies the above before consent, they will be excluded from the trial
      * They will also be excluded from the trial if they have suffered any fractured bones in the last 3 months (this will further decrease risk to the patient as the patient will be moved by the physician during the treatment protocol)
      * Participants who are enrolled in other Long-COVID trials that have an intervention during their participation in this trial will be excluded. However, if they have a history of enrollment in a long-covid trial that has no interventions during this trial, they will not be excluded based on their history of acquiring experimental treatment.

      IV: Statistical Analysis Plan:

      The data acquired from the SBQ™-LC will be used to determine changes in long covid symptom burden and change relative to treatment participant received. As of right now, the team has secured the licensure to use the physical paper SBQ™-LC; there are current attempts to acquire a digital version to help assist with logistics and bring down burden on the research participants relative to data collection. All participants will take the survey a total of 4 times, the first being administered on arrival and consenting process as a baseline followed by one administered every 7 days. The survey will be uploaded via RedCap and sent to participants electronically.

      The SBQ™-LC has n=123 symptoms in 17 different scales measured with the target population being Adults (18+ years) living with post-COVID condition, also known as post-acute sequelae of COVID-19 (PASC), or Long COVID. In addition, the fact that there are multiple different scales within the SBQ™-LC, there can be analysis based on this treatment efficacy based on different symptom constellations. For example: this treatment may only be helpful for olfactory function and not gastro-intestinal symptoms, this survey will help differentiate this question.

      There will be one experimental group to control group survey that will give info on benefit of one vs no treatment. Then there will be a 2 consecutive treatment group to 1 treatment comparison. This will help identify if participants benefit from multiple treatments or if only one treatment is enough for symptom management as well as assist with assessing the placebo effect.

      Finally, BP and HR will be acquired for participants while in the clinic. This will give us proxy information to see if there is an impact on this treatment relative to participants sympathetic tone.

      Statistical Analysis: Continuous variables will be summarized using mean and standard deviation if they are normally distributed or using median and interquartile range if they are not normally distributed. The Smirnov-Kolmogorov test will be used to evaluate normality. Categorical variables will be summarized with frequency count and percentage. Linear mixed models will be used to evaluate the change pre-post treatment in symptoms' scores as well as the difference of that change between different groups. The mixed models will include a group variable (with 2 categories: OMT, sham), a timepoint variable (pre-post treatment), and their intersection. Random intercept and slope will be included for each participant to account for individual variability and change. Linear contrasts will be built on the interaction term to obtain estimates of different comparisons for the study. All tests will be 2-sided. The significance level will be set to 5%. If the linear model assumptions are not satisfied, variable transformations will be explored. To account for multiple comparisons, the p-values will be adjusted accordingly using Bonferroni correction or similar methods, and care will be taken in the interpretation of the results.

      Power Analysis: In the analysis, the pre-post treatment changes will be compared between the treatment group (OMT) and the sham group. In the pilot study, we have observed an effect of OMT of effect sizes of 0.63-1.9. We would like to detect the median of those effect sizes, 1.2 classified as huge on the Sawilowsky's extension of Cohen criteria. Group sample sizes of 8 for OMT and 8 for sham achieve over 80% power to detect this effect size using a 2-sided Mann-Whitney U test assuming a double exponential data distribution of the data (a conservative option) with a significance level of 0.05. To account for potential loss of data, we will enroll 20% participants in each group, i.e. 10 participants per group for a total of 20.

      IVa. Risks to patients:

      - Lightheadedness/dizziness post-treatment

      - Drowsiness post-treatment

      - Potential frustration related to no improvement of symptoms

      IVb. Risk Mitigation system:

      - There will be a 10-minute timer after each treatment before vitals are assessed.

      - Participants will be asked to report any side effects

      - All adverse events will be recorded and submitted to University of Louisville IRB in concordance with IRB adverse event identification protocol.

      IVc. Good Clinical Practices and Good Laboratory Practices All participants will have adequate time to be consented as well as ask any questions regarding the project. University of Louisville IRB approval will be completed prior to initiating the research. Participants will be made aware of all side effects prior to treatment. All participants will be made aware that participation in this trial is voluntary and they can exit the trial at any time.

      IVd. Discussion of major anticipated challenges:

      The largest challenge in this study will be maintaining follow up with these participants. The research team will generate an electronic SBQ™-LC survey to make participant participation have a higher likelihood of completion due to decreased physical logistical burden.

      V Informed Consent Process:

      Consent will be obtained upon participant physical arrival to the study site. Consent documents will be given to participant prior to any survey distribution or vital signs acquirement. After consent is obtained, participant will begin survey prior to vital signs or treatment is initiated. An approved study team member will be acquiring consent for all participants.

      Citations

      [1] Mollica V, Rizzo A, Massari F. The pivotal role of TMPRSS2 in coronavirus disease 2019 and prostate cancer. Future Oncol. 2020;16(27):2029-2033. doi:10.2217/fon-2020-0571

      [2] Gengler, I, Wang, JC, Speth, MM, Sedaghat, AR. Sinonasal pathophysiology of SARS-CoV-2 and COVID-19: A systematic review of the current evidence. Laryngoscope Investigative Otolaryngology. 2020; 5: 354- 359. https://doi.org/10.1002/lio2.384

      [3] Butowt R, von Bartheld CS. Anosmia in COVID-19: Underlying Mechanisms and Assessment of an Olfactory Route to Brain Infection [published online ahead of print, 2020 Sep 11]. Neuroscientist. 2020;1073858420956905. doi:10.1177/1073858420956905

      [4] Lechien, Jerome R et al. "Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study." European archives of oto-rhino-laryngology: official journal of the European Federation of Oto-Rhino-Laryngological Societies (EUFOS): affiliated with the German Society for Oto-Rhino-Laryng

      [5] Bryche B, St Albin A, Murri S, et al. Massive transient damage of the olfactory epithelium associated with infection of sustentacular cells by SARS-CoV-2 in golden Syrian hamsters. Brain Behav Immun. 2020;89:579-586. doi:10.1016/j.bbi.2020.06.032

      [6] Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc. 2005 Oct;105(10):447-56. PMID: 16314677.

      [7] Hughes SE, Haroon S, Subramanian A, McMullan C, Aiyegbusi OL, Turner GM, Jackson L, Davies EH, Frost C, McNamara G, Price G, Matthews K, Camaradou J, Ormerod J, Walker A, Calvert MJ. Development and validation of the symptom burden questionnaire for long covid (SBQ-LC): Rasch analysis. BMJ. 2022 Apr 27;377:e070230. doi: 10.1136/bmj-2022-070230.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals must claim they have had a prior positive SARS-CoV-2 test at least 6-weeks before the consenting process to proceed with the study
* Individuals must claim they have at least one of the following symptoms greater than 6-weeks post infection that is affecting their daily life(these symptoms correlate with the SBQ™-LC):

Symptoms of Long Covid Inclusion Criteria:

* Shortness of breath or Difficulty Breathing
* Difficulty with Movement (balance or tremor)
* Muscle Pain or stiffness
* Changes in sexual desire
* Worsening Generalized Pain
* Difficulty with Sleep
* Changes in Mood (anxiety or depression)
* Changes in Erectile function (Biological males only)
* Palpations (irregular heart beats)
* Altered Taste
* Changes in your Hair
* Changes in urination
* Dizziness
* Altered Smell
* Changes in Skin
* Changes in bowels
* Fatigue
* Indigestion
* Dry or irritated eyes
* Changes in sweating
* Difficulty with Cognition (memory or thinking)
* Stomach Pain
* Changes in menstruation (Biological females only)
* Chills or shivering

Exclusion Criteria:

* If anyone denies they have any of the above symptoms before consent, they will be excluded from the trial

  * They will also be excluded from the trial if they have suffered any fractured bones in the last 3 months (this will further decrease risk to the patient as the patient will be moved by the physician during the treatment protocol)
  * Participants who are enrolled in other Long-COVID trials that have an intervention during their participation in this trial will be excluded. However, if they have a history of enrollment in a long-covid trial that has no interventions during this trial, they will not be excluded based on their history of acquiring experimental treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
The Symptom Burden Questionnaire™ for Long COVID (SBQ™-LC) | On arrival for baseline before any treatment (week 1). On arrival for 2nd treatment (week 2). 7 days after 2nd treatment (week 3). Final Survey on week 8 of post-enrollment
  The Symptom Burden Questionnaire™ for Long COVID (SBQ™-LC) is a validated tool generated to assess for Long-COVID symptom burden generated by the University of Birmingham in the UK. The SBQ™-LC assesses 123 different symptoms of Long COVID.
  All items use the recall period "In the last 7 days..." and are scored according to one of the following:
  1. symptom presence (Yes/No);
  2. symptom frequency (0 = Never to 3 = Always);
  3. symptom severity (0 = None to 3 = Severe);
  4. or Interference in daily life (0 = Not at all to 3 = Severely). The SBQ™-LC has a Flesch-Kincaid Reading Grade level score of 5.33 suggesting it would be understood by a person with a 6th grade reading level according to the American education system. The SBQ™-LC's SMOG Index score of 8.27 means it should be understood by 93% of UK adults.(8-10)
  Higher scores suggest worsening symptom severity.
  Maximum raw score depends on which independent scale within the tool is measured. Ranges from 5-38 depending

SECONDARY OUTCOMES:
Blood Pressure(BP) | Each in-person treatment event, total of 1 BP at arrival after being enrolled for baseline and then a repeat 10 minutes after treatment (regardless of which treatment arm); repeat sequence at the 2nd in-person visit for a total of 4 BP readings
  BP's will be taken before treatment regardless of arm participants are assigned at baseline. It will be repeated 10 minutes after the each treatment
Heart Rate (HR) | Each in-person treatment event, total of 1 HR at arrival after being enrolled for baseline and then a repeat 10 minutes after treatment (regardless of which treatment arm); repeat sequence at the 2nd in-person visit for a total of 4 HR readings
  HR's will be taken before treatment regardless of arm participants are assigned at baseline. It will be repeated 10 minutes after the each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Kaelin, MD, Medical Doctorate (US), Principal Investigator — University of Louisville School of Medicine Chair of PM&R Division of the Department of Neurological Surgery
Locations (1):
- University of Louisville Outpatient Care Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Study protocol, Statistical analysis plan will be shared during journal submission

REFERENCES:
- [Background] Hughes SE, Haroon S, Subramanian A, McMullan C, Aiyegbusi OL, Turner GM, Jackson L, Davies EH, Frost C, McNamara G, Price G, Matthews K, Camaradou J, Ormerod J, Walker A, Calvert MJ. Development and validation of the symptom burden questionnaire for long covid (SBQ-LC): Rasch analysis. BMJ. 2022 Apr 27;377:e070230. doi: 10.1136/bmj-2022-070230. PMID 35477524
- [Background] Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc. 2005 Oct;105(10):447-56. PMID 16314677
- [Background] Bryche B, St Albin A, Murri S, Lacote S, Pulido C, Ar Gouilh M, Lesellier S, Servat A, Wasniewski M, Picard-Meyer E, Monchatre-Leroy E, Volmer R, Rampin O, Le Goffic R, Marianneau P, Meunier N. Massive transient damage of the olfactory epithelium associated with infection of sustentacular cells by SARS-CoV-2 in golden Syrian hamsters. Brain Behav Immun. 2020 Oct;89:579-586. doi: 10.1016/j.bbi.2020.06.032. Epub 2020 Jul 3. PMID 32629042
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Butowt R, von Bartheld CS. Anosmia in COVID-19: Underlying Mechanisms and Assessment of an Olfactory Route to Brain Infection. Neuroscientist. 2021 Dec;27(6):582-603. doi: 10.1177/1073858420956905. Epub 2020 Sep 11. PMID 32914699
- [Background] Gengler I, Wang JC, Speth MM, Sedaghat AR. Sinonasal pathophysiology of SARS-CoV-2 and COVID-19: A systematic review of the current evidence. Laryngoscope Investig Otolaryngol. 2020 Apr 16;5(3):354-359. doi: 10.1002/lio2.384. eCollection 2020 Jun. PMID 32587887
- [Background] Mollica V, Rizzo A, Massari F. The pivotal role of TMPRSS2 in coronavirus disease 2019 and prostate cancer. Future Oncol. 2020 Sep;16(27):2029-2033. doi: 10.2217/fon-2020-0571. Epub 2020 Jul 13. No abstract available. PMID 32658591